CLINICAL TRIAL: NCT06324110
Title: Evaluating Centralizing Interventions to Address Low Adherence to Lung Cancer Screening Follow-Up in Decentralized Settings (The ACCELL Interventional Trial)
Brief Title: Evaluating the Impact of Centralized Interventions on Lung Cancer Screening Adherence in Community Settings, ACCELL Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RG1124119; NCI-2024-01763 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20250 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA284032 (NIH)
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Interviews as Topic; Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (LCS coordination) (Experimental): Patients receive lung cancer screening follow-up care coordination services, delivered by a lung cancer screening care coordinator at their care site.
  Interventions: Other: Electronic Health Record Review; Other: Interview; Behavioral: Patient Navigation

INTERVENTIONS:
Other: Electronic Health Record Review — Ancillary studies
Other: Interview — Ancillary studies
Behavioral: Patient Navigation — Receive lung cancer screening care coordination services
  Other Names: Patient Navigator Program

SUMMARY:
This clinical trial tests the impact of lung cancer screening care coordination interventions implemented at the system-level on lung cancer screening adherence in community settings. Lung cancer remains the leading cause of cancer death in the United States. Although lung cancer screening (LCS) with yearly low-dose chest computed tomography has the potential to decrease lung deaths, the use of this screening technique remains low. In addition, studies have shown that adherence to lung cancer screening in clinical settings is far lower that those found in clinical trials. Improved care coordination services that include comprehensive, system-wide tracking of screening outcomes for all LCS participants, results reporting with direct-to-patient information, direct patient and physician communication, and active reviews of non-adherent patients and stepped support interventions may increase patient adherence to LCS. Coordination services at the system-level may decrease barriers and improve adherence to lung cancer screening in community settings.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive lung cancer screening follow-up care coordination services, delivered by a lung cancer screening care coordinator at their care site.

ELIGIBILITY:
Inclusion Criteria:

* AIM II: Age 50-80
* AIM II: Current or former (within 15 years) smoker
* AIM II: 20+ pack-years of cigarette use
* AIM II: Undergone at least one lung cancer screening low-dose chest computed tomography (CT) at partnering sites within the study period
* AIM III (PROVIDER INTERVIEWS): Age minimum of 18
* AIM III (PROVIDER INTERVIEWS): Affiliation with Skagit Regional Health System, Confluence Health or Kadlec Regional Medical Center
* AIM III (PROVIDER INTERVIEWS): Identifies as providing primary care or specialty care to LCS patients (medical doctor [MD], registered nurse [RN], physician assistant [PA], advanced registered nurse practitioner [ARNP])
* AIM III (LCS PATIENT INTERVIEWS): Aged 50-80 years
* AIM III (LCS PATIENT INTERVIEWS): Received lung cancer screening at Skagit Regional Health System, Confluence Health or Kadlec Regional Medical Center within the intervention period
* AIM III (LCS PATIENT INTERVIEWS): Was eligible for LCS at time of performance by United States Preventative Services Taskforce (USPSTF) criteria

  * Age 50-80 at time of exam
  * At least 20 pack-year smoking history
  * Currently smoking or smoked within the last 15 years
* AIM III (LCS-SPECIFIC CARE COORDINATORS): Age minimum of 18
* AIM III (LCS-SPECIFIC CARE COORDINATORS): Affiliation with Skagit Regional Health System, Confluence Health or Kadlec Regional Medical Center
* AIM III (LCS-SPECIFIC CARE COORDINATORS): Identifies as fulfilling a supportive role in the LCS care continuum as part of the centralizing intervention

Exclusion Criteria:

* AIM II: No longer eligible for lung cancer screening chest CT during follow-up period (no longer meeting inclusion criteria during follow-up period)
* AIM II: Request to not participate in the trial
* AIM III (PROVIDER INTERVIEWS): Less than age 18
* AIM III (PROVIDER INTERVIEWS): Do not have an affiliation with Skagit Regional Health System, Confluence Health or Kadlec Regional Medical Center
* AIM III (PROVIDER INTERVIEWS): Does not identify as providing primary care or specialty care to LCS patients (MD, RN, PA, ARNP)
* AIM III (LCS PATIENT INTERVIEWS): Less than age 50 or older than age 80
* AIM III (LCS PATIENT INTERVIEWS): Did not receive lung cancer screening at Skagit Regional Health System, Confluence Health or Kadlec Regional Medical Center within the intervention period
* AIM III (LCS PATIENT INTERVIEWS): Was not eligible for LCS at time of performance by USPSTF criteria
* AIM III (LCS-SPECIFIC CARE COORDINATORS): Less than of 18
* AIM III (LCS-SPECIFIC CARE COORDINATORS): Does not have an affiliation with Skagit Regional Health System, Confluence Health or Kadlec Regional Medical Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6772 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to appropriate follow-up | Up to 48 months
  The time and covariate adjusted difference in adherence to appropriate follow-up will be assessed between the pre- and post-intervention period, separately for negative and positive exams. Follow-up will be considered on-time if occurring by the recommended follow up window + 30 days. The impact of the interventions on follow-up will be measured a using generalized estimating equations (GEE)-based approach. The modeling will be done using logistic regression. The Bonferroni correction will be used to account for testing two intervention coefficients.

SECONDARY OUTCOMES:
Characteristics associated with adherence to follow up | Up to 48 months
  The impact of site, patient race/ethnicity, socioeconomic status and patient rurality on adherence will be evaluated in both the pre-intervention and the post-intervention period. The impact of site and patient characteristics on the pre-intervention adherence rate will be evaluated with multivariable logistic regression models using GEE to account for multiple rounds of lung cancer screening within an individual patient. Associations of site and patient characteristics with extent of delay for non-adherent patients will be evaluated using multivariable accelerated failure time models. The overall follow-up rate will be analyzed using multivariable Cox regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Triplette, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Louie T, Snidarich M, Hippe DS, Wernli KJ, Palazzo L, Hansell L, Brown M, Coronado GD, Lodhi S, Leone R, DeCell K, Mardesich K, Wysham N, Triplette M. A pragmatic pre-post intervention trial to address adherence to lung cancer screening follow-up in community settings (the ACCELL trial): Study protocol. Contemp Clin Trials. 2025 Dec;159:108106. doi: 10.1016/j.cct.2025.108106. Epub 2025 Oct 10. PMID 41076116